CLINICAL TRIAL: NCT05178043
Title: A Phase II Study to Evaluate the Efficacy and Safety of GT90001 in Combination With Nivolumab as a Second-line Treatment in Subjects With Advanced Hepatocellular Carcinoma
Brief Title: GT90001 Plus Nivolumab in Patients With Advanced Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GT90001-MR-1001
Record Dates: First submitted 2021-11-25; First posted 2022-01-05 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab; ascrinvacumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GT90001+Nivolumab (Experimental)
  Interventions: Drug: Nivolumab; Drug: GT90001

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 240mg to be administered as an intravenous (IV) infusion every 2 weeks (Q2W).
  Other Names: Opdivo, ONO-4538, BMS-936558, MDX1106
Drug: GT90001 — GT90001 7mg/kg to be administered as an intravenous infusion every 2 weeks (Q2W) after Nivolumab infusion.
  Other Names: PF-03446962

SUMMARY:
This is a global phase II, open label study in the subjects with Advanced Hepatocellular Carcinoma (aHCC) who were intolerant or had progressed after or intolerant to first-line Immune Checkpoint Inhibitors (ICI) such as Atezolizumab plus Bevacizumab, or ICI plus Tyrosine Kinase Inhibitor (TKI).

Based on published and first-hand experience with the safety and tolerability of both GT90001 and Nivolumab, the proposed dose is GT90001 7 mg/kg in combination with Nivolumab 240 mg, infusion every two weeks.

This study will enroll a total of 105 subjects to receive combinational therapy of Nivolumab and GT90001.

• Nivolumab 240 mg will first be administered by intravenous infusion over 30 minutes, then 30 minutes later, give intravenous infusion of GT90001 7.0 mg/kg over 60 min, once every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have confirmed diagnosis of aHCC (locally advanced or metastatic hepatocellular carcinoma) by radiography, histology and/or cytology, not eligible for surgical and/or locoregional therapies; or progressive disease after surgical and/or locoregional therapies (fibrolamellar, sarcomatoid HCC and mixed hepatocellular / cholangiocarcinoma subtypes are not eligible);
* Have Barcelona Clinic Liver Cancer (BCLC) Stage C disease or BCLC Stage B disease not amenable to locoregional therapy or refractory to locoregional therapy;
* Have documented disease progression after or intolerance to first line treatment of immune checkpoint inhibitors(ICI)
* Child-Pugh score ≤ 6 (Child-Pugh A) score within 7 days of first dose of study drug;
* ECOG performance status: 0-1 within 7 days of first dose of study drug;
* Have a predicted life expectancy of greater than 3 months;
* Adequate hematologic and end-organ function functions of the important organs are confirmed.

Exclusion Criteria:

* Presence of tumor thrombus involving main trunk of portal vein (Vp4), inferior vena cava, cardiac involvement of HCC;
* Subjects with untreated or incompletely treated varices with bleeding or high-risk for bleeding. Has had esophageal or gastric variceal bleeding within the last 6 months;
* History of encephalopathy;
* Has a known history of, or any evidence of central nervous system (CNS) metastases and/or carcinomatous meningitis;
* Had history of a solid organ or hematologic transplant;
* Has received locoregional therapy to liver (TACE, TAE, hepatic arterial infusion [HAI], radiation, radioembolization or ablation) within 4 weeks of start of study treatment.
* Had prior systemic TKI treatment prior to start of study treatment;
* Has received prior immune checkpoint inhibitors within 4 weeks of start of study treatment;
* Has received Nivolumab in the first-line systemic therapy:
* Active co-infection with:

  1. Both hepatitis B and C as evidenced by positive HBV surface antigen or detectable HBV DNA and HCV RNA, OR
  2. Hepatitis D infection in subjects with hepatitis B
* Has an active bacterial or fungal infection requiring systemic therapy within 7 days prior to study drug dosing;
* Has a known history of active tuberculosis (Bacillus Tuberculosis);
* Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture;
* Thrombotic or embolic events (except HCC tumor thrombus) within the past 6 months, such as cerebrovascular accident (including transient ischemic attacks), pulmonary embolism; If prior history of deep vein thrombosis (DVT) / (pulmonary embolism (PE), the subject needs to be on stable doses of anticoagulation with low molecular weight heparin or oral anticoagulant for at least two weeks;
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis;
* Subjects with any other serious disease considered by the investigator not in the condition to enter into the trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The Objective Response Rate (ORR) (confirmed) as evaluated by an Independent Review Committee (IRC) according to RECIST v1.1 | Approximately 2 years
  ORR is defined as the proportion of participants with best overall response of confirmed complete response (CR) or partial response (PR). RECIST: Response Evaluation Criteria in Solid Tumors

SECONDARY OUTCOMES:
Duration OF Response (DOR) as evaluated by an IRC according to RECIST v1.1 | Approximately 2 years
Progression Free Survival (PFS) as evaluated by an IRC according to RECIST v1.1 | Approximately 2 years
Time To Response (TTR) as evaluated by an IRC according to RECIST v1.1 | Approximately 2 years
Time to Progression (TTP) as evaluated by an IRC according to RECIST v1.1 | Approximately 2 years
Disease Control Rate (DCR) as evaluated by an IRC according to RECIST v1.1 | Approximately 2 years
ORR (confirmed) as evaluated by the investigator according to RECIST v1.1 | Approximately 2 years
DOR as evaluated by the investigator according to RECIST v1.1 | Approximately 2 years
PFS as evaluated by the investigator according to RECIST v1.1 | Approximately 2 years
TTR as evaluated by the investigator according to RECIST v1.1 | Approximately 2 years
TTP as evaluated by the investigator according to RECIST v1.1 | Approximately 2 years
DCR as evaluated by the investigator according to RECIST v1.1 | Approximately 2 years
ORR (confirmed) as evaluated by an IRC according to HCC mRECIST | Approximately 2 years
DOR as evaluated by an IRC according to HCC mRECIST | Approximately 2 years
PFS as evaluated by an IRC according to HCC mRECIST | Approximately 2 years
TTR as evaluated by an IRC according to HCC mRECIST | Approximately 2 years
TTP as evaluated by an IRC according to HCC mRECIST | Approximately 2 years
DCR as evaluated by an IRC according to HCC mRECIST | Approximately 2 years
ORR (confirmed) as evaluated by the investigator according to HCC mRECIST | Approximately 2 years
DOR as evaluated by the investigator according to HCC mRECIST | Approximately 2 years
PFS as evaluated by the investigator according to HCC mRECIST | Approximately 2 years
TTR as evaluated by the investigator according to HCC mRECIST | Approximately 2 years
TTP as evaluated by the investigator according to HCC mRECIST | Approximately 2 years
DCR as evaluated by the investigator according to HCC mRECIST | Approximately 2 years
Overall survival (OS) | Approximately 3 years
Safety and tolerability (any Advense Events (AEs), Severe AEs , immune-related AEs (irAEs), treatment-related AEs, abnormal laboratory values, etc. | Approximately 2 years
Presence of Anti-Drug Antibodies (ADAs) to GT90001 and Nivolumab during the study relative to the presence of ADAs at baseline | Approximately 2 years

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - City of Hope National Medical Center, Duarte, California
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - NYU Langone Health, New York, New York
  - Renovatio Clinical, Houston, Texas
  - Medical Oncology Associates, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided